CLINICAL TRIAL: NCT05912413
Title: Prediction of Sepsis Recovery Physical Performance Subtypes: A Pilot Study
Brief Title: Predicton of Sepsis Recovery Performance Subtypes Pilot Study
Status: Recruiting | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Peter Morris, Professor, University of Alabama at Birmingham
Other Study IDs: IRB-300010502-003
Record Dates: First submitted 2023-06-02; First posted 2023-06-22 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: there is no intervention — there is no intervention

SUMMARY:
This study addresses critically ill sepsis patients' current literature reports of ongoing post-hospital discharge weakness and hospital readmissions. This study is aimed at capture and interpretation of a complex set of tests, administered during a subject's sepsis functional recovery trajectory, particularly capturing hospital readmission's effects on survivors' physical function recovery.

DETAILED DESCRIPTION:
Patients with Sepsis who require ICU care, experience frequent weakness, physical dysfunction, fatigue, difficulty concentrating, poor memory, and mental morbidity that persists after hospital discharge. This syndromic pattern has been labeled as Post Intensive Care Syndrome (PICS) or Post Sepsis Syndrome (PSS). These patients are at increased risk of rehospitalization (up to 40% at 6 months). Studies have pointed out that sepsis survivors recover within several different recovery patterns or trajectories. Unfortunately there are no objective biomarkers early in these patients' hospitalizations, to predict which physical function trajectory a sepsis survivor will experience. However, a very common, unifying symptom of sepsis survivors is weakness. The literature maintains that an intervention of exercise rehabilitation remains a safe and potential therapy for sepsis survivors. It is important to note that as of yet, there has been no benefit demonstrated when highly heterogeneously functioning survivors are included in studies of a uniform rehabilitation intervention. However, for the future designs of ICU and post-hospital ICU Survivor exercise-rehab trials, the field is in need of information on how to label sepsis patients by their predicted outpatient recovery trajectory group, and to be able to do so very proximally in their course, prior to hospital discharge. The intent of this study is to closely track and characterize physical function recovery trajectory groups as a means of informing strategies for effective future study design.

ELIGIBILITY:
Inclusion Criteria:

* Sepsis requiring organ support in an ICU setting

Exclusion Criteria:

1. inability to obtain informed consent
2. the attending physician reports that the patient's goals of care are transitioning to palliation/withdrawal of life-sustaining therapy
3. recent cancer therapy in the last 12 months
4. age >80
5. plans to be discharged on mechanical ventilation to a Long Term Acute Care Hospital
6. planned discharge to rehabilitation facility, long-term hospital or nursing home.
7. Pregnancy

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Sepsis requiring organ support in an ICU setting
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-07-11 (Actual); Primary Completion 2025-10-15 (Estimated); Study Completion 2025-10-15 (Estimated)

PRIMARY OUTCOMES:
Short Performance Physical Battery | 3 months post hospital discharge
  Physical function score

CONTACTS AND LOCATIONS:
Overall Officials: peter morris, md, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham (UAB) Hospital, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Undecided
undecided